CLINICAL TRIAL: NCT02902913
Title: Impact of Extra Virgin Olive Oil Oleocanthal Content on Platelet Reactivity in Healthy Humans
Brief Title: Impact of Extra Virgin Olive Oil Oleocanthal Content on Platelet Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 617247
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Results first posted 2019-11-07 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases
Keywords: platelet reactivity; phenolic; extra virgin olive oil; cyclooxygenase; oleocanthal; oxylipin
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: All participants received all four interventions in a randomized, cross-over design in which both participant and caregiver were masked to the assignment (with the exception of the fourth intervention, ibuprofen, which was always administered at the final study visit).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oleocanthal-rich, D2i2 (Experimental): Oleocanthal-rich, D2i2 (Extra virgin olive oil containing oleocanthal to oleacein in a 2:1 ratio)
  Interventions: Other: D2i2
- Oleacein-rich, D2i0.5 (Experimental): Oleacein-rich, D2i0.5 (Extra virgin olive oil containing oleocanthal to oleacein in a 1:2 ratio)
  Interventions: Other: D2i0.5
- Oleocanthal and Oleacein-low, D2i0 (Placebo Comparator): Oleocanthal and Oleacein-low, D2i0 (Extra virgin olive oil containing low amounts of oleocanthal to oleacein, but with a similar total phenolic content as the other two oils)
  Interventions: Other: D2i0
- Ibuprofen (Active Comparator): Ibuprofen, 400 mg
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Other: D2i2 — Oleocanthal provided in a 2:1 ratio compared to oleacein
  Other Names: Oleocanthal-rich
  Arms: Oleocanthal-rich, D2i2
Other: D2i0.5 — Oleocanthal provided in a 1:2 ratio compared to oleacein
  Other Names: Oleocanthal-low
  Arms: Oleacein-rich, D2i0.5
Other: D2i0 — No oleocanthal and no oleacein
  Other Names: Control EVOO
  Arms: Oleocanthal and Oleacein-low, D2i0
Drug: Ibuprofen — 400 mg of Ibuprofen
  Arms: Ibuprofen

SUMMARY:
Data from limited dietary intervention trials suggest that the cardiovascular health benefit of extra virgin olive oil (EVOO) may increase with phenolic content. However, while EVOOs contain an array of bioactive compounds, little information exists regarding the physiological effects of specific chemical species. Among the EVOO-derived phenolics with demonstrated anti-inflammatory effects in animal and in vitro models is oleocanthal, an inhibitor of cyclooxygenase (COX). The current study compared the impact of acute intake (40 mL) of EVOO on platelet reactivity in healthy adult males (n=9). The volunteers were randomly assigned to consume three EVOOs in a double-blind controlled trial. The EVOO were characterized and chosen for equivalency in their total phenolic content and fatty acid profiles, but differing in their oleocanthal to oleacein ratio.

DETAILED DESCRIPTION:
Ten healthy adult males (20-50 years of age) will be enrolled into a randomized triple-blind, controlled crossover study that will test the acute effects of oleocanthal-rich extra virgin olive oil intake on platelet aggregation. Each participant will be asked to participate in four study days, separated by at least 1-week, in which they will be randomized to consume on each study day 40 mL (~3 tablespoons) of either oleocanthal-rich extra virgin olive oil (OO), or an extra virgin OO that is matched in total phenolics but oleocanthal-poor, or a refined OO that is low in all phenolics In addition to the oils, on a fourth study day visit, after completion of the study visits involving oil intake the subjects will be asked to take 400mg of ibuprofen.

Collection procedures will be performed at the same time of the day to avoid circadian effects. A blood sample (50 mL ~ 3.5 tbsp) will be collected for the measurement of platelet aggregometry and COX metabolites. Following this initial blood draw, the subjects will consume their assigned test product for the day. Two-hours following the intake of the assigned olive oil, a second blood sample will be drawn (50 mL ~ 3.5 tbsp). After the second blood draw, the study day will be complete.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with study protocols
* Willing to drink 2 tablespoons of olive oil
* BMI 18.5 to 30 kg/m2
* Weight ≥ 110 pounds

Exclusion Criteria:

* Adults who are not able to consent
* BMI ≥ 31 kg/m2
* Under current medical supervision
* Self-reported daily use of drugs that are known to affect platelet function, such as aspirin, Excedrin, and NSAIDS
* Ibuprofen intolerance or allergy
* Cannot speak English
* Allergy to olives or olive oil
* Vegetarian, Vegan, food faddists, individuals using non-traditional diets, on a weight loss diet or individual following diets with significant deviations from the average diet of the general population.
* A history of cardiovascular disease, stroke, cancer, renal, hepatic, or thyroid disease, GI tract disorders, previous GI surgery
* Currently taking prescription drugs or supplements
* Indications of substance or alcohol abuse within the last 3 years
* Not willing to stop any supplement use, including herbal, plant or botanical, fish oil, oil supplements.
* Not willing to refrain from olive oil consumption.
* Blood Pressure ≥ 140/90 mmHg
* Self-reported malabsorption
* Metabolic panel results or complete blood counts that are outside of the normal reference range.
* Screening LDL ≥ 190 mg/dl for those who have 0 - 1 major risk factors apart from LDL cholesterol [(i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL].
* Screening LDL ≥ 160 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [(i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL].
* Screening LDL ≥ than 130 mg/dl for those who have 2 major risk factors apart from LDL cholesterol ((i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL), and a Framingham 10 - year Risk Score 10 - 20 % (using NCEP calculator).
* Current enrollee in a clinical research study.
* Individuals with blood clotting or platelet defect disorders

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta R Holt, PhD, Principal Investigator — University of California, Davis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Agrawal K, Melliou E, Li X, Pedersen TL, Wang SC, Magiatis P, Newman JW, Holt RR. Oleocanthal-rich extra virgin olive oil demonstrates acute anti-platelet effects in healthy men in a randomized trial. J Funct Foods. 2017 Sep;36:84-93. doi: 10.1016/j.jff.2017.06.046. Epub 2017 Jul 3. PMID 29904393
- See also: manuscript — https://pubmed.ncbi.nlm.nih.gov/29904393/

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants received all four study interventions. The first three interventions were administered in random order:
  * Oleocanthal-rich, D2i2
  * Oleacein-rich, D2i0.5
  * Oleocanthal and Oleacein-low, D2i0
  All participants received the last intervention, 400 mg of Ibuprofen, at the fourth (final) study visit.
Period: Overall Study
Arm/Group | All Participants
Started | 9
First Intervention (1 Day) | 9
Washout (7 Days) | 9
Second Intervention (1 Day) | 9
Washout (7 Days) | 9
Third Intervention (1 Day) | 9
Washout (7 Days) | 9
Ibuprofen (400mg) | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Optical Platelet Aggregometry
Description: Maximal platelet aggregation in minutes will be measured using optical platelet aggregometry
Time Frame: Change from baseline 2 hours post intake
Measure: Mean (Standard Deviation); unit: percentage of maximal aggregation
Arm/Group | All Participants
Number analyzed (Participants) | 9
percentage of maximal aggregation
  D2i2 | -13 (36)
  D2i0.5 | -35 (39)
  D2i0 | 7 (24)
  Ibuprofen | -57.5 (32.9)

2. Secondary Outcome: Activated Platelet Oxylipin Production
Description: Oxylipins derived from cyclooxygenase, lipoxygenase, and cytochrome P450 dependent metabolism of AA were quantified using liquid chromatography with tandem mass spectrometry (LC-MS/MS) in 100 µL of PRP plasma activated with collagen or ADP as well as 100 µL of unactivated PRP plasma collected before and two hours after treatment with EVOO or ibuprofen.
  Data were mean centered and reported as a % change from baseline.
Time Frame: Change from baseline 2 hours post intake
Population: healthy adult males
Measure: Number; unit: percentage of change from baseline
Arm/Group | Oleocanthal-rich, D2i2 | Oleacein-rich, D2i0.5 | Oleocanthal and Oleacein-low, D2i0 | Ibuprofen
Number analyzed (Participants) | 9 | 9 | 9 | 9
percentage of change from baseline | -0.02 | -0.45 | -0.17 | -0.66

ADVERSE EVENTS:
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No